CLINICAL TRIAL: NCT00132184
Title: Remission Keeping and Remission Inducing Effect by Vitamin-D in Crohns Disease, and in Vitro Vitamin-D Mediated T-Cell Immunomodulation
Brief Title: Vitamin D Treatment for Crohn´s Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-001216-50
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2007-04-13 (Estimated); Status verified 2007-04

CONDITIONS: Crohns Disease
Keywords: Vitamin D; Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
The purpose of this study is to examine whether vitamin D treatment is effective in Crohn's disease.

DETAILED DESCRIPTION:
Crohns Disease is an inflammatory disease of primarily the small intestine and colon.

In recent years scientists have hypothesized that low blood vitamin-D levels play a role in the development of autoimmune diseases, including Crohns disease. The purpose of this study is to examine whether vitamin-D is effective in keeping remission in inactive Crohns Disease (double blind placebo controlled trial). The patients who have active disease in the placebo group (reach primary endpoint), will in an open setting receive a higher single dose vitamin-D and the effect will be measured within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease
* Inactive Crohn's disease for at least 4 weeks
* Crohn's Disease Activity Index (CDAI) < 150
* C-reactive protein within normal range
* Serum albumin within normal range

Exclusion Criteria:

* Hypercalcemia
* Short bowel syndrome
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2005-09; Study Completion 2008-02 (Estimated)

PRIMARY OUTCOMES:
Relapse rate within 1 year treatment; CDAI>220

CONTACTS AND LOCATIONS:
Overall Officials: Jens F. Dahlerup, MD, DrMedSc, Principal Investigator — Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Aarhus University Hospital, Department V, Aarhus
  - Hospital of Horsens, Horsens
  - Hospital of Randers, Randers
  - Hospital of Silkeborg, Silkeborg